CLINICAL TRIAL: NCT02494921
Title: A Phase 1b/2 Study of the Oral CDK4/6 Inhibitor LEE011 (Ribociclib) in Combination With Docetaxel Plus Prednisone in Metastatic Castration Resistant Prostate Cancer
Brief Title: LEE011 (Ribociclib) in Combination With Docetaxel Plus Prednisone in mCRPC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 145515; NCI-2015-01797 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; ribociclib; Prednisone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Phase 1b) (Experimental): The starting cohort dose level (1) for docetaxel will be 75 mg/m2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily, starting on day 1 of the 21-day cycle. If dose level 1 is not tolerated, then alternative dosing schedules of docetaxel will be evaluated, starting with dose level 1A of 60mg/m2 docetaxel.
  Interventions: Drug: Docetaxel-PNP; Drug: Ribociclib; Drug: Prednisone; Drug: Filgrastim
- Treatment (Phase 2) (Experimental): Participants in Phase 2 will receive the Recommended Phase 2 Dose for docetaxel and ribociclib
  Interventions: Drug: Docetaxel-PNP; Drug: Ribociclib; Drug: Prednisone; Drug: Filgrastim

INTERVENTIONS:
Drug: Docetaxel-PNP — Given IV
  Other Names: Taxotere; Docetaxel Injection
Drug: Ribociclib — Given Orally
  Other Names: Kisqali
Drug: Prednisone — Given Orally
  Other Names: Prednisone Oral
Drug: Filgrastim — Given IV
  Other Names: Neupogen

SUMMARY:
This is a Phase Ib/II open label clinical trial in patients with metastatic castration resistant prostate cancer. The objective of the phase Ib portion of the study is to establish the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of docetaxel (75 mg/m2 IV q21 days) and prednisone (5mg orally BID) in combination with ribociclib in escalating oral daily doses in patients with metastatic castrate resistant prostate cancer (mCRPC) with prior resistance to abiraterone and/or enzalutamide who have not undergone prior chemotherapy for metastatic disease. Up to three cohorts will be enrolled to determine the MTD and DLT profile of this combination during Phase 1b. Dose escalation will follow the standard 3+3 design. The dosing schedule is being chosen to allow patients to be exposed to the most efficacious dosing schedule of docetaxel (75 mg/m2 every 3 weeks). If there is excess toxicity observed with the treatment combination at the first dose level (dose level I), an alternative dosing schema may be pursued with weekly docetaxel treatment (35 mg/m2 weekly), which has demonstrated activity in mCRPC and decreased risk of cytopenias compared with every 3 week dosing schedule.

The Phase II portion (N = 29) of the study is a single arm, two stage, open-label study of ribociclib (dosed at the RP2D) in combination with docetaxel and prednisone to determine the efficacy and further define the safety of the treatment combination. Patients will be treated with the combination of ribociclib plus docetaxel + prednisone for up to 9 cycles. If there is no evidence of radiographic or clinical disease progression after 9 cycles of protocol therapy, patients may continue on single agent maintenance ribociclib until the time of disease progression. Patients will have the option of starting maintenance ribociclib after 6 cycles of docetaxel if stable disease or better on re-staging scans. The dose of ribociclib used during maintenance will be the same dose as that immediately preceding cessation of docetaxel treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile, maximally tolerated dose (MTD), and recommended phase 2 dose of ribociclib in combination with docetaxel plus prednisone in patients with metastatic castration-resistant prostate cancer (mCRPC). (Phase IB) II. To determine the 6-month radiographic progression-free survival rate with the combination of ribociclib, docetaxel, and prednisone in patients with mCRPC. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the median radiographic progression-free survival with the combination of ribociclib, docetaxel, and prednisone in patients with mCRPC.

II. To determine the objective response rate and median duration of response among patients with measurable disease at baseline.

III. To determine the prostate-specific antigen (PSA) response proportion and time to PSA progression.

IV. To characterize the safety profile of ribociclib in combination with docetaxel.

V. To determine if there is evidence of drug-drug interaction between docetaxel + prednisone with ribociclib.

EXPLORATORY OBJECTIVES:

I. To determine whether baseline or percent change from baseline in gallium citrate uptake on positron emission tomography (PET) scan is associated with clinical outcomes. (For University of California San Francisco (USCF) Patients Only) II. To determine whether genomic assessment of MYC pathway activation (MYC amplification or overexpression, Rb1 deletion, cyclin D/E and CDK 4/6 overexpression) assessed within metastatic tumor tissue, circulating tumor cells (CTCs), and/or cell-free circulating tumor deoxyribonucleic acid (ctDNA) is predictive of clinical outcomes with the combination of ribociclib plus docetaxel.

III. To determine whether MYC activation score as determined by validated expression signature can distinguish those with and without clinical benefit with ribociclib in combination with docetaxel.

IV. To use an unbiased approach with integration of clinical, genomic, and proteomic data (differential pathway signature correlation; DiPSC) to define a signature associated with response to taxane + CDK4/6 inhibition in mCRPC.

OUTLINE: This is a phase Ib, dose-escalation study of ribociclib followed by a phase II study.

Patients receive docetaxel intravenously (IV) over 1 hour on day 1 or on days 1 and 8, prednisone orally (PO) twice daily (BID) on days 1-21, and ribociclib PO once daily (QD) on days 1-4, and 8-15. Treatment repeats every 21 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better on re-staging scans after 6 cycles and patients without radiographic or clinical disease progression after 9 cycles of treatment may continue on single agent maintenance ribociclib PO QD on days 1-14 of every 21 day cycle in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every three months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer. Small cell/neuroendocrine differentiated allowed but not required for study participation.
* Progressive metastatic prostate cancer (as defined below in Item #5) despite castrate levels of testosterone (< 50 ng/dL).
* Patients may have either non-measurable disease OR measurable disease
* Progressive disease during (or within 4 weeks of completion) with abiraterone, enzalutamide, and/or ARN-509 based on any one of the following:

  1. For patients with measurable disease, progression by the RECIST criteria.
  2. PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least one week apart. If the confirmatory PSA (#3) value is less (i.e., #3b) than the screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression for the purposes of eligibility.
  3. Radionuclide bone scan: At least two new foci consistent with metastatic lesions
* Testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with a luteinizing hormone-releasing hormone (LHRH) analogue if they have not undergone orchiectomy.
* Patients treated with first generation anti-androgen as most recent systemic therapy (bicalutamide, nilutamide) must have at least 4 weeks elapsed from treatment discontinuation to start of protocol therapy with evidence of disease progression by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria following discontinuation of prior anti-androgen.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:
* Absolute neutrophil count ≥ 1.5 × 109/L.
* Platelets ≥ 100 × 109/L.
* Hemoglobin ≥ 9 g/dl.
* Potassium, total calcium (corrected for serum albumin) and magnesium within normal limits for the institution or corrected to within normal limits before first dose of study medication.
* International normalized ratio (INR) ≤ 1.5 unless on direct thrombin inhibitor at time of study entry.
* Serum creatinine ≤ 1.5mg/dL or estimated creatinine clearance ≥ 50 ml/min
* In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x upper limit of normal (ULN). If the patient has liver metastases, ALT and AST <5 x ULN
* Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
* No other systemic therapies for prostate cancer within 28 days or 5 half-lives, whichever is shorter, prior to day 1 of study therapy.
* Sexually active males must use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. Fertile males must use a condom with spermicide (double barrier method).
* Age ≥ 18 years
* Written informed consent must be obtained prior to any screening procedures and according to local guidelines.

Exclusion Criteria:

* Patient has a known hypersensitivity to ribociclib or any of its excipients, or prior treatment with cyclin-dependent kinase (CDK) 4/6 inhibitor.
* Prior chemotherapy for metastatic castration-resistant prostate cancer. Chemotherapy administered in the castration-sensitive setting is allowed provided last dose of chemotherapy was greater than 6 months prior to study entry
* Patient has a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated, basal cell skin cancer, squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Patients with central nervous system (CNS) involvement unless they meet all of the following criteria:
* At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
* Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* Baseline screening for CNS metastases is not required unless presence of signs and/or symptoms of involvement
* Patient is not able to swallow oral medication and/or has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or significant small bowel resection).
* Clinically significant, uncontrolled heart disease and/or recent events including any of the following:
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 12 months prior to screening
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Patient has a left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) obtained during Screening.
* History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening. Patients with rate-controlled atrial fibrillation or flutter are permitted.
* Bradycardia (heart rate < 50 bpm at rest), by ECG or pulse, at screening
* Congenital long QT syndrome or family history of long QT syndrome
* Any of the following abnormalities on screening 12-lead ECG:
* QT interval with Fridericia's correction (QTcF) > 450 msec
* Bradycardia (heart rate < 50 bpm at rest)
* Tachycardia (heart rate > 100 bpm at rest)
* P-R interval > 220msec,
* QRS interval >109 msec
* Documented cardiomyopathy
* Systolic blood pressure >160 mmHg or <90 mmHg at screening
* AST and/or ALT > 1.5 x ULN with concomitant alkaline phosphatase > 2.5 x ULN
* Patient receiving any of the following medications within 7 days of day 1 of study treatment.
* Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
* That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
* That have a known risk to prolong the QT interval or induce Torsades de Pointes.
* Herbal preparations/medications
* Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug at a dose greater than the equivalent of 10 mg prednisone/day, or who have not fully recovered from the side effects of such treatment
* The following uses of corticosteroids are permitted: short duration (<5 days) of systemic corticosteroids; any duration of topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, direct thrombin inhibitors, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
* Major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia), and/or in whom ≥25% of the bone marrow was irradiated.
* Patient has a known history of HIV infection (testing not required)
* Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 to less than or equal to Grade 1 (Exception to this criterion: patients with grade 1 taxane-induced neuropathy, any grade of alopecia, amenorrhea or other toxicities not considered a safety risk for the patient as per investigator's discretion, are allowed to enter the study).
* Patients with chronic liver disease with a Child-Pugh score B or C.
* Patients with serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
* Patients with severe psychiatric illness/social situations that would limit compliance with study requirements in the judgment of study investigator.
* History of bleeding diathesis. Patients receiving anti-coagulation must be able safely interrupt treatment for tumor biopsy (Phase 2 only)
* Patient has a history of non-compliance to medical regimen or inability to grant consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial dosing schedule was chosen as the most efficacious dosing schedule of docetaxel. If dose level I is not tolerated, then alternative dosing schedules of docetaxel were evaluated, starting with dose level IA. Depending on the safety data observed, alternative dosing schedules and intermediate dose levels of ribociclib was investigated (Cohort / Dose Levels IC - IIIC) per protocol.
Groups:
- Treatment (Phase 1b, Non-RP2D, Cohort I): The starting cohort dose level (1) for docetaxel will be 75 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily, starting on day 1 of the 21-day cycle.
- Treatment (Phase 1b, Non-RP2D, Cohort IA): The starting cohort dose level (1) for docetaxel will be 60 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily, starting on day 1 of the 21-day cycle.
- Treatment (Phase 1b, Non-RP2D, Cohort IIC): The starting cohort dose level (1) for docetaxel will be 60 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 300 mg orally once daily, starting on day 1 of the 21-day cycle.
- Treatment (Phase 1b, R2PD, Cohort IIIC); Treatment (Phase 2, RP2D): The starting cohort dose level (1) for docetaxel will be 60 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 400 mg orally once daily, starting on day 1 of the 21-day cycle.
Period: Phase 1b, Dose Level I
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Started | 5 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Period: Phase 1b, Dose Level IA
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Started | 0 | 4 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Phase 1b, Dose Level IIC
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Started | 0 | 0 | 4 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Period: Phase 1b, Dose Level IIIC, RP2D
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Started | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase 2, RP2D
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Started | 0 | 0 | 0 | 0 | 24
Completed | 0 | 0 | 0 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants assigned to the recommended phase 2 dose (RP2D) during their Phase 1b enrollment, were included in the Phase 1b/2 RP2D group for data analysis
Groups:
- Treatment (Phase 1b, RP2D, Cohort IIIC); Treatment (Phase 2, RP2D): The starting cohort dose level (1) for docetaxel will be 60 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 400 mg orally once daily, starting on day 1 of the 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, RP2D, Cohort IIIC) | Treatment (Phase 2, RP2D) | Total
Number analyzed (Participants) | 5 | 4 | 4 | 6 | 24 | 43
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 3 | 0 | 0 | 1 | 1 | 5
  60-69 years | 1 | 1 | 2 | 3 | 13 | 20
  70-79 years | 1 | 2 | 2 | 2 | 9 | 16
  80-89 years | 0 | 1 | 0 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 4 | 4 | 6 | 24 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 1 | 4
  Not Hispanic or Latino | 5 | 2 | 3 | 5 | 22 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 4 | 4 | 4 | 4 | 19 | 35
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 6 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) (Phase 1b)
Description: Maximally tolerated dose (MTD) of ribociclib in combination with docetaxel and prednisone is based upon evaluation of dose-limiting toxicities (DLTs) and adverse events for all participants who received treatment in Phase Ib. If 1 of 3 participants in a cohort experiences a DLT, then the cohort will be expanded to treat an additional 3 participants. If only 1 of 6 participants experiences a DLT, the next cohort of participants will be treated at the next higher dose level. If 2 or more participants in a cohort experience a DLT, then MTD has been exceeded and the previous dose level will be considered the MTD. If more than 1 of 6 patients experience a DLT at dose level IA then the study will be terminated, as the MTD cannot be determined and de-escalation from dose level IA is not planned. Per Investigator discretion the Recommended Phase 2 Dose (RP2D) schedule of ribociclib and docetaxel may be established in the absence of reaching MTD.
Time Frame: Up to 2 years
Population: All participants in Phase 1b including those who received the RP2D were included in this analysis
Measure: Number; unit: mg/m^2
Groups:
- Treatment (Phase 1b): The starting cohort dose level (I) for docetaxel will be 75 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily, starting on day 1 of the 21-day cycle. If dose level (1) is not tolerated, then alternative dosing schedules of docetaxel will be evaluated, starting with dose level IA of 60mg/m2 docetaxel.
Arm/Group | Treatment (Phase 1b)
Number analyzed (Participants) | 19
mg/m^2 | NA — MTD was not reached

2. Primary Outcome: RP2D of Docetaxel (Phase 1b)
Description: The RP2D of docetaxel will be reported when used in combination with ribociclib and prednisone based upon evaluation of dose-limiting toxicities (DLTs) and adverse events for all participants in the Phase Ib group. Per Investigator discretion, the RP2D schedule of docetaxel and ribociclib may be established in the absence of reaching MTD, based on the cumulative safety data of the treatment regimen.
Time Frame: Up to 2 years
Population: All participants in Phase 1b, including those who received the Recommended Phase 2 Dose for docetaxel and ribociclib will be included in the analysis. The final RP2D was determined to be 60mg/m^2 of docetaxel in combination with 400mg of ribociclib.
Measure: Number; unit: mg/m^2
Groups:
- Treatment (Phase 1b): The starting cohort dose level (1) for docetaxel will be 75 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily, starting on day 1 of the 21-day cycle. If dose level 1 is not tolerated, then alternative dosing schedules of docetaxel will be evaluated, starting with dose level 1A of 60mg/m2 docetaxel.
Arm/Group | Treatment (Phase 1b)
Number analyzed (Participants) | 19
mg/m^2 | 60

3. Primary Outcome: Percentage of Participants With Radiographic Progression-free Survival at 6 Months (Phase 1b/2 RP2D)
Description: Radiographic progression-free survival will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percent of participants has been estimated using the Kaplan-Meier product limit method. Duration will be measured from day 1 of study treatment to first date of radiographic progression or death, whichever occurs first, for all Phase 1b or Phase 2 participants receiving the RP2D. Participants who discontinue study therapy for toxicity, withdrawal from study, or prostate-specific antigen (PSA)-only progression, will be censored at the date of last radiographic tumor assessment for this analysis. Patients who discontinue therapy for evidence of clinical progression/clinical deterioration will be included in this analysis.
Time Frame: Up to 6 months
Population: All participants in Phase 1b (N=6) and Phase 2 (N=24) who received the RP2D were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Phase 1b/2 RP2D): Participants in Phase 1b and Phase 2 who received the Recommended Phase 2 Dose for docetaxel and ribociclib.
Arm/Group | Treatment (Phase 1b/2 RP2D)
Number analyzed (Participants) | 30
percentage of participants | 65.8 [50.6 to 85.5]

4. Secondary Outcome: Median Radiographic Progression-free Survival (Phase1b/2 RP2D)
Description: Radiographic progression-free survival will be assessed using RECIST version 1.1. Median duration will be Estimated using the Kaplan-Meier product limit method. Duration will be measured from day 1 of study treatment to first date of radiographic progression or death, whichever occurs sooner for participants in Phase 1b and Phase 2 who receive the RP2D. Participants who discontinue study therapy for toxicity, withdrawal from study, or prostate-specific antigen (PSA)-only progression, will be censored at the date of last radiographic tumor assessment for this analysis. Participants who discontinue therapy for evidence of clinical progression/clinical deterioration will be included in this analysis.
Time Frame: Up to 2 years
Population: All participants in Phase 1b (N=6) and Phase 2 (N=24) who received the RP2D were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Phase 1b/2 RP2D)
Number analyzed (Participants) | 30
months | 8.09 [6.89 to 10.03]

5. Secondary Outcome: Objective Response Rate (ORR) (Phase1b/2 RP2D)
Description: ORR will be assessed using RECIST version 1.1 criteria, and defined as participants who were determined to have demonstrated a complete response (CR) and/or partial response (PR). Participants must have measurable disease at baseline with at least one restaging scan on treatment to be included in the analysis.
Time Frame: Up to 2 years
Population: Of 30 possible participants, only 13 met the criteria of both measurable disease at baseline and at least one restaging scan on treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Phase 1b/2 RP2D)
Number analyzed (Participants) | 13
percentage of participants | 23.1 [9.1 to 61.4]

6. Secondary Outcome: Median Duration of Response (Phase1b/2 RP2D)
Description: For participants with both measurable disease at baseline and at least one restaging scan on treatment, duration of response will be defined as the time criteria are met for CR or PR until recurrent or progressive disease is objectively documented.
Time Frame: Up to 2 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Treatment (Phase 1b/2): Participants in Phase 1b and Phase 2 who received the Recommended Phase 2 Dose for docetaxel and ribociclib.
Arm/Group | Treatment (Phase 1b/2)
Number analyzed (Participants) | 13
days | 141.5 [59 to 259]

7. Secondary Outcome: Prostate-Specific Antigen (PSA) Response Rate (Phase 1b/2 RP2D)
Description: PSA progression occurs when the PSA value has increased 25% or greater above nadir and an absolute increase of 2 ng/mL or more from the nadir is documented. Where no decline is observed, PSA progression similarly occurs when a 25% increase from baseline value along with an increase in absolute value of 2 ng/mL or more per the Prostate Cancer Working Group 2 (PCWG2) Criteria.
Time Frame: Up to 2 years
Population: Of 30 possible participants, 5 participants did not have documented PSA response values available and were excluded from the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Phase 1b/2 RP2D)
Number analyzed (Participants) | 25
percentage of participants | 32 [15.0 to 53.5]

8. Secondary Outcome: Median PSA Progression-Free Survival (Phase 1b/2 RP2D)
Description: The PSA response duration commences on the date of the first 50% decline in PSA. The response duration ends when the PSA value increases by 25% above the nadir, provided that the increase in the absolute-value PSA level is at least 5 ng/mL or back to baseline, whichever is lower. The probability distribution of the median time to PSA progression will be estimated using the Kaplan-Meier product limit method.
Time Frame: Up to 2 years
Population: Of 30 possible participants, 8 participants were excluded from the analysis due to lack of documented PSA after baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Phase 1b/2 RP2D)
Number analyzed (Participants) | 22
months | 7.15 [2.86 to 8.45]

9. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: The number of participants with reported adverse events related to the treatment regimen will be descriptively reported using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Analyses will be performed for all patients having received at least one dose of study drug.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, R2PD, Cohort IIIC) | Treatment (Phase 2, RP2D)
Number analyzed (Participants) | 5 | 4 | 4 | 6 | 24
Participants | 5 | 4 | 4 | 6 | 22

10. Secondary Outcome: Mean Area Under Curve (AUC) 0-24 Hour (Phase 1b)
Description: The estimated AUC for serum concentration of ribociclib for a 24 hour interval after dose will be reported using descriptive statistics for all participants in Phase 1b who received at least one dose of study treatment and completed a serum blood draw.
Time Frame: Pre-dose on day 1, and 1, 2, 4, and 24 hours post-dose
Population: All participants in Phase 1b, Non-RP2D were grouped for this analysis since the drug of interest is ribociclib only. All participants in the combined Phase 1b, non-RP2D group did not receive the 400 mg dose at any time, and 1 participant did not have serum levels recorded. Participants in the combined Phase 1b, RP2D cohort did not receive < 400 mg dose at any time.
Measure: Mean (95% Confidence Interval); unit: ng*hrs/mL
Groups:
- Treatment (Phase 1b, Non-RP2D): The starting cohort dose level (1) for docetaxel will be 75 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 200 mg orally once daily and increase to 300mg for additional cohorts if tolerated, starting on day 1 of the 21-day cycle. If dose level 1 is not tolerated, then alternative dosing schedules of docetaxel will be evaluated, starting with dose level 1A of 60mg/m^2 docetaxel.
- Treatment (Phase 1b, RP2D): The starting cohort dose level (1) for docetaxel will be 60 mg/m^2, administered on day 1 of each cycle. Prednisone will be fixed at 5 mg twice a day. The starting dose level and schedule for ribociclib will begin at 400 mg orally once daily, starting on day 1 of the 21-day cycle.
Arm/Group | Treatment (Phase 1b, Non-RP2D) | Treatment (Phase 1b, RP2D)
Number analyzed (Participants) | 12 | 6
ng*hrs/mL
  200 mg ribociclib: number analyzed (Participants) | 9 | 0
  200 mg ribociclib | 2909 [1699.7 to 4119.2] |
  300 mg ribociclib: number analyzed (Participants) | 3 | 0
  300 mg ribociclib | 3340.3 [1825.3 to 6491.1] |
  400 mg ribociclib: number analyzed (Participants) | 0 | 6
  400 mg ribociclib |  | 6531.6 [2922.5 to 10140.6]

11. Secondary Outcome: Mean Maximum Serum Concentration of Ribociclib (Cmax) (Phase 1b)
Description: The maximum concentration (Cmax) is shown to reflect not only the rate but also the extent of absorption. The mean Cmax for serum concentration of ribociclib will be reported using descriptive statistics for all participants in Phase 1b who received at least one dose of study treatment and completed a serum blood draw.
Time Frame: Pre-dose on day 1, and 1, 2, 4, and 24 hours post-dose
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment (Phase 1b, Non-RP2D) | Treatment (Phase 1b, RP2D)
Number analyzed (Participants) | 12 | 6
ng/mL
  200 mg Ribociclib: number analyzed (Participants) | 9 | 0
  200 mg Ribociclib | 207.5 [135.4 to 279.6] |
  300 mg Ribociclib: number analyzed (Participants) | 3 | 0
  300 mg Ribociclib | 289.8 [92.5 to 672] |
  400 mg Ribociclib: number analyzed (Participants) | 0 | 6
  400 mg Ribociclib |  | 393.6 [139.5 to 647.6]

12. Secondary Outcome: Estimated Steady-state Serum Concentration (Csteady-state) (Phase 1b)
Description: Steady-state serum concentration occurs when the amount of a drug being absorbed is the same amount that is being cleared from the body when the drug is given continuously. Steady-state concentration is the time during which the concentration of the drug in the body stays consistent. The estimated steady state for serum concentration of ribociclib will be reported using descriptive statistics for all participants in Phase 1b who received a steady dosing schedule of study treatment and completed a serum blood draw.
Time Frame: Up to 2 years
Population: An intermittent ribociclib dosing scheduled was pursued so a steady-state serum concentration level could not be determined.
Arm/Group | Treatment (Phase 1b, Non-RP2D) | Treatment (Phase 1b, RP2D)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Phase 1b, Non-RP2D, Cohort I) | Treatment (Phase 1b, Non-RP2D, Cohort IA) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) | Treatment (Phase 1b, RP2D, Cohort IIIC) | Treatment (Phase 2, RP2D)
All-Cause Mortality (participants affected / at risk) | 4/5 | 1/4 | 3/4 | 3/6 | 11/24
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/4 | 0/4 | 3/6 | 5/24
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 4/4 | 6/6 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Phase 1b, Non-RP2D, Cohort I) (N=5) | Treatment (Phase 1b, Non-RP2D, Cohort IA) (N=4) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) (N=4) | Treatment (Phase 1b, RP2D, Cohort IIIC) (N=6) | Treatment (Phase 2, RP2D) (N=24)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right lower visual field cut (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Phase 1b, Non-RP2D, Cohort I) (N=5) | Treatment (Phase 1b, Non-RP2D, Cohort IA) (N=4) | Treatment (Phase 1b, Non-RP2D, Cohort IIC) (N=4) | Treatment (Phase 1b, RP2D, Cohort IIIC) (N=6) | Treatment (Phase 2, RP2D) (N=24)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0) | 3 (5) | 5 (8)
Hypoprotenemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypertension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (intermittent) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epiphoria (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (6) | 10 (19)
Bilateral hip pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilateral posterior rib pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone and hand discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (7)
Fatigue (General disorders) | 3 (3) | 3 (3) | 2 (3) | 5 (11) | 14 (20)
Fever (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left anterolateral rib pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left pubic rami pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neck edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Sleep disturbances (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (6) | 1 (1)
International Normalized Ratio (INR) increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (12)
Neutrophil count decreased (Investigations) | 4 (16) | 3 (7) | 1 (1) | 3 (5) | 10 (19)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
White blood cell decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) — Muscle cramps
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Muscle aches
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) — Joint aches
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (5)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 7 (7)
Light headedness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 9 (9)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Chest Congestion
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 8 (9)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Nail changes
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Pruritic Rash
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Phosphorous (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders, Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) — Muscle Spasms

LIMITATIONS AND CAVEATS:
Participants assigned to the Phase 1b RP2D cohort were included in a combined Phase 1b/2 RP2D group for some of the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02494921/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT02494921/ICF_001.pdf